CLINICAL TRIAL: NCT02237560
Title: The Cognitive Benefits of Interactive Mental and Physical Exercise for Older Adults at Risk for or With Mild Cognitive Impairment (MCI)
Brief Title: The Aerobic & Cognitive Exercise Study
Acronym: ACES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Union College, New York (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Cay Anderson-Hanley, PhD, Associate Professor, Union College, New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS13083; R15AG042109-01A1 (NIH)
Record Dates: First submitted 2014-09-04; First posted 2014-09-11 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Mild Cognitive Impairment; Healthy
Keywords: MCI; Exergaming; Cognition; Exercise; Older Adults
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cybercycle-Game (Experimental): Combined aerobic & cognitive exercise for 6 months, 3-5x/week.
  Interventions: Behavioral: Cybercycle-Game
- Cybercyle-Tour (Active Comparator): Aerobic exercise only for 6 months, 3-5x/week.
  Interventions: Behavioral: Cybercyle-Tour
- Game Only (Active Comparator): Cognitive exercise only 6 months, 3-5x/week.
  Interventions: Behavioral: Game Only

INTERVENTIONS:
Behavioral: Cybercycle-Game — Exercising on a virtual-reality enhanced stationary recumbent bicycle while playing interactive 3D video-game for 6 months, 3-5x/week.
  Other Names: Expresso; Dragon Chase
  Arms: Cybercycle-Game
Behavioral: Cybercyle-Tour — Exercising on virtual-reality enhanced stationary recumbent bicycle and pedaling through interactive 3D scenic bike tours for 6 months, 3-5x/week.
  Other Names: Expresso
  Arms: Cybercyle-Tour
Behavioral: Game Only — While seated on a stationary recumbent seat play interactive 3D video-game for 6 months, 3-5x/week (no pedaling).
  Other Names: Dragon Chase
  Arms: Game Only

SUMMARY:
The purpose of this study is to clarify the benefits to brain health and thinking processes that result from different forms of exercise. This study will examine the effectiveness of cybercycling (virtual reality enhanced stationary cycling) for persons at risk for and with MCI, and compare this with the individual cognitive, behavioral, and physiological effects of physical and mental exercise alone. The Investigators hypothesis that cognitive benefit will be greatest for combined aerobic and cognitive exercise compared to physical and mental exercise alone.

DETAILED DESCRIPTION:
This is a multi-site, randomized controlled trial. Participants will be randomized into one of three conditions for six months: cybercycle-tour, cybercycle-game, or videogame alone. Comprehensive evaluations will include: neuropsychological (e.g., executive function and memory), behavioral (e.g., compliance and effort/watts), physiological (e.g., cardiorespiratory fitness), biomarker (e.g., BDNF), and an expanded neuroimaging pilot. After the six-month intervention period, participants choose whether or not to continue exercising, using any of the three conditions.

ELIGIBILITY:
Inclusion Criteria:

* age 50+
* able to pedal recumbent stationary bicycle
* available for regular exercise participation 3-5x/week for at least 6 months
* physician permission to exercise

Exclusion Criteria:

* unstable heart condition or other significant cardiovascular history (e.g,. stroke)
* meets criteria for Alzheimer's or other dementia
* significant history of other neurological disease (e.g., seizures, Parkinson's, etc.)
* physician denial to exercise

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2014-09; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in executive function at 6-months | Baseline and 6-months
  Change in executive function from baseline at 6-months will be assessed by using a composite executive function score obtained from scores on Digit Span Backwards, Stroop, and Color Trails.

SECONDARY OUTCOMES:
Change in weight | Baseline, 3-months, 6-months, 1-year
  Weight and other physiological factors will be assessed at baseline, 3-months, 6-months, and 1-year follow-up
Change in mood | Baseline, 3-months, 6-months, 1-year follow-up
  Behavioral outcomes (e.g., mood) will be assessed using the Brunel Mood Scale and exercise induced feeling inventory.
Change from baseline in executive function at 3-months | Baseline and 3-months
  Change from baseline in executive function will be assessed using composite executive function score obtained from scores on Digit Span Backwards, Stroop, and Color Trails.
Change from baseline in executive function at 1-year follow-up | Baseline and 1-year
  Change from baseline in executive function will be assessed using composite executive function score obtained from scores on Digit Span Backwards, Stroop, and Color Trails.

OTHER OUTCOMES:
Change from baseline in BDNF at 6-months | Baseline and 6-months
  BDNF levels (collected from saliva samples) at 6-months will be compared with baseline levels.
Change from baseline in MRI at 6-months | Baseline and 6-months
  MRI scans collected at baseline and 6-months will be analyzed for volumetric changes.
Cognitive characteristics of sample pre- and post- intervention | Baseline and 6-months
  The MoCA, ADAS-Cog word recall, complex figures, and controlled oral word association test will be used to characterize the sample based on cognitive function at pre- and post-intervention.
Assessment of exercise behavior during intervention | After each exercise session
  Participants are asked to exercise 3-5x/week. After each exercise session subjects will record their exercise data (e.g., time, distance, power, heart rate, calories, points).

CONTACTS AND LOCATIONS:
Overall Officials: Cay Anderson-Hanley, PhD, Principal Investigator — Union College
Locations (12):
- United States (12):
  - Albany Medical Center, Albany, New York
  - Sidney Albert Albany Jewish Community Center, Albany, New York
  - Stratton VA Medical Center, Albany, New York
  - Hawthorne Ridge, East Greenbush, New York
  - Guilderland YMCA, Guilderland, New York
  - Glen Eddy, Niskayuna, New York
  - Coburg Village, Rexford, New York
  - Prestwick Chase, Saratoga Springs, New York
  - Kingsway Parkland GardenApartments, Schenectady, New York
  - Schaffer Heights, Schenectady, New York
  - Sunnyview Rehabilitation Center, Schenectady, New York
  - Beverwyck, Slingerlands, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anderson-Hanley C, Barcelos NM, Zimmerman EA, Gillen RW, Dunnam M, Cohen BD, Yerokhin V, Miller KE, Hayes DJ, Arciero PJ, Maloney M, Kramer AF. The Aerobic and Cognitive Exercise Study (ACES) for Community-Dwelling Older Adults With or At-Risk for Mild Cognitive Impairment (MCI): Neuropsychological, Neurobiological and Neuroimaging Outcomes of a Randomized Clinical Trial. Front Aging Neurosci. 2018 May 4;10:76. doi: 10.3389/fnagi.2018.00076. eCollection 2018. PMID 29780318